CLINICAL TRIAL: NCT04416828
Title: Medical Imaging in the Diagnosis of Ganglion Cysts of the Hand
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Waldfriede Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019.4
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Ganglion Cyst of Both Hands
Keywords: Portable ultrasound; Diagnostics; Mobile ultrasound; Hand held ultrasound; Wireless ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected ganglion cyst of the wrist or hand: Patients with suspected ganglion cyst of the wrist or hand receive portable wireless ultrasound imaging AND cart-based ultrasound imaging before surgery.
  Interventions: Device: Portable wireless ultrasonography devices; Device: Cart-based ultrasonography device

INTERVENTIONS:
Device: Portable wireless ultrasonography devices — Patients with suspected ganglion cyst of the wrist or hand receive portable wireless ultrasound imaging
Device: Cart-based ultrasonography device — Patients with suspected ganglion cyst of the wrist or hand receive conventional cart-based ultrasound imaging

SUMMARY:
The aim of this study is to investigate if inexpensive, readily available and portable wireless ultrasound devices can detect ganglion cysts of the wrist and hand in compare to a cart-based ultrasound device before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Flexor tendon sheath ganglion cyst
* Dorsal ganglion cyst
* Palmar ganglion cyst
* Male and female patients minimum age 18 years
* MRI of the affected area

Exclusion Criteria:

* Pregnancy, lactation
* Malignant disease
* Insufficient mental possibility of cooperation
* Medical, psychiatric or other conditions that restrict the patient's following abilities: to interpret the study information, to give informed consent, to adhere to the rules of the protocol, or to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ninety male and female patients with ganglion cyst of the wrist or hand planned for surgery will be recruited at the hand surgery outpatient clinic of the Waldfriede Hospital Berlin. Patients will be diagnosed with ganglion cyst of the hand/wrist by an experienced hand surgeon using clinical and MRI data.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-06-04 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Size and location of ganglion cysts of the wrist and hand | Baseline (pre-surgery)
  Assessment of size in cm and location of the ganglion cyst of the wrist or hand by pre-surgery wireless ultrasound in compare to pre-surgery cart-based ultrasound

SECONDARY OUTCOMES:
MRI measure of size and location of ganglion cysts of the wrist and hand | Baseline (pre-surgery)
  Assessment of size in cm and location of the ganglion cyst of the wrist or hand by pre-surgery MRI in compare to pre-surgery ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lautenbach, MD, Study Chair — Hospital Waldfriede, Argentinische Allee 40, 14163 Berlin; Markus Bock, MD, Principal Investigator — Hospital Waldfriede, Argentinische Allee 40, 14163 Berlin
Locations (1):
- Waldfriede Hospital, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No